CLINICAL TRIAL: NCT05846724
Title: A Phase II Single-arm Study of Pembrolizumab Plus Lenvatinib in Previously Treated Classic Kaposi Sarcoma (CKS)
Brief Title: Pembrolizumab Plus Lenvatinib in Previously Treated Classic Kaposi Sarcoma
Acronym: PULSAR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The lack of adequate funding has made it impossible to continue with the clinical study As this study was not initiated, no subject was included and no data was collected,thus no result can be obtained SPONSOR_DECISION End of trial date:15 Oct 2025
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-3475-B60
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2023-01

CONDITIONS: Kaposi Sarcoma; Classic Kaposi Sarcoma; Refractory Kaposi Sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Pembrolizumab + Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab + Lenvatinib — single-arm study of pembrolizumab plus lenvatinib

SUMMARY:
Phase II study of Pembrolizumab plus Lenvatinib in relapsed/refractory Classic Kaposi Sarcoma (CKS). After a screening phase of up to 28 days, each participant will receive study intervention of pembrolizumab plus lenvatinib until reaching a discontinuation criterion: disease progression; unacceptable adverse event(s) (AEs); intercurrent illness that prevents further administration of treatment; participant withdraws consent; pregnancy of participant; non-compliance with study intervention or procedure requirements; or administrative reasons requiring cessation of treatment.

After the end of treatment, each participant will be followed for the occurrence of AEs and spontaneously reported pregnancy.

Participants who discontinue for reasons other than PD will have post-treatment follow-up for disease status until PD is documented clinically by a team of committed dermatologists, and/or radiographically per RECIST 1.1, a non-study anticancer treatment is initiated, consent is withdrawn, or the participant becomes lost to follow-up.

All participants will be followed for overall survival (OS) until death, withdrawal of consent,lost to follow-up, or the end of the study. The end of the study will be when the last participant completes the last study-related telephone call or visit,withdraws from the study, or is lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically confirmed diagnosis of classic (or endemic) KS
2. Progression or inadequate response to at least one prior systemic chemotherapy
3. Presence of measurable disease by PET-CT scan and/or dermatological examination
4. KS with at least 10 cutaneous and/or mucosal lesions, or involving more than one limb segment or with involvement >3% body surface
5. KS with at least 4 lesions ≥ 5mm
6. KS with at least 1 superficial lesion willing to provide tissue from cutaneous and/or mucosal biopsy at baseline
7. At least 4 weeks washout for all KS specific therapies including chemotherapy (both systemic and intralesional) and radiotherapy
8. Be ≥ 18 years of age at the time of signing informed consent
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
10. Have adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg and no change in antihypertensive medications within 1 week prior to randomization.

Exclusion Criteria:

1. Has a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies detected at screening).
2. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
3. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with vitiligo, type I diabetes mellitus, hypothyroidism, psoriasis not requiring systemic treatment are permitted to enroll.
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
5. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) of pembrolizumab with lenvatinib in pre-treated recurrent CKS | 6 months
  the combination of pembrolizumab and lenvatinib has superior ORR, as compared to cytotoxic chemotherapy by literature data. ORR defined as a confirmed complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Duration of response (DOR) in patients with pre-treated recurrent CKS receiving pembrolizumab with lenvatinib | 6 months
  The combination of pembrolizumab and lenvatinib provides superior DOR, as compared to cytotoxic chemotherapy by literature data.
Progression Free Survival (PFS) of patients with pre-treated recurrent CKS receiving pembrolizumab with lenvatinib. | 6 months
  The combination of pembrolizumab and lenvatinib has superior PFS, as compared to cytotoxic chemotherapy by literature data.
Overall Survival in patients receiving pembrolizumab and lenvatinib | 6 months
  The combination of pembrolizumab and lenvatinib has superior OS, as compared to cytotoxic chemotherapy by literature data.
The mean change from baseline in the global health status/quality of life (QoL), and physical functioning for the combinations of pembrolizumab and lenvatinib | 6 months
  Score for the following patient-reported outcomes (PROs) scales/items: global health status/QoL (EORTC QLQ-C30items 29 and 30), and physical functioning (EORTC QLQ-C30 items 1-5).
Safety and tolerability for the combination of pembrolizumab and lenvatinib. | 6 months
  Adverse Events (AEs) incidence and study intervention discontinuation due to AEs